CLINICAL TRIAL: NCT01875744
Title: Polyethylene Glycol for Childhood Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Andrea Horvath-Stolarczyk, MD PhD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 2/2013; 2/2013 (Other Grant/Funding Number: The Medical University of Warsaw)
Record Dates: First submitted 2013-06-06; First posted 2013-06-12 (Estimated); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Constipation
Keywords: constipation; children; polyethylene glycol
MeSH Terms: conditions — Constipation | interventions — polyethylene glycol 4000

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyethylene glycol small dose (Experimental): Polyethylene glycol 4000: 0.3 g/kg/day for 6 weeks
  Interventions: Drug: Polyethylene glycol 4000
- Polyethylene glycol high dose (Active Comparator): Polyethylene glycol 4000: 0.7g/kg for 6 weeks
  Interventions: Drug: Polyethylene glycol 4000

INTERVENTIONS:
Drug: Polyethylene glycol 4000
  Other Names: Forlax

SUMMARY:
Background:

Aim:

Clinical evaluation of the effectiveness of two different polyethylene glycol doses for the maintenance treatment of functional constipation in children.

Study design:

Randomized, open-label trial.

Randomized, double-blind, placebo controlled trial.

DETAILED DESCRIPTION:
Children will be randomly assigned into 2 groups receiving polyethylene glycol 4000 (Forlax) with an initial dose of either 0.3g/kg, or 0.7 g / kg.

In case of ineffectiveness the dose of medication will be increased every two weeks with 0.2 g/kg. The indication for the increase in dose will be less than 3 bowel movements per week. For children with diarrhea defined as more than 3 loose stools for minimum 2 days or/and severe abdominal pain the macrogol dose of will be reduced every two weeks by 0.2 g/kg. The intervention will last 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age 1 - 18 age
* functional constipation according to the Rome III Criteria
* consent of parents or guardians of the child to participate and study

Exclusion Criteria:

* organic cause constipation (including surgeries within the lower GI tract)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11-30 (Actual)

PRIMARY OUTCOMES:
therapeutic success (passing ≥ 3 stools per week, with no loosening of stool). | the number and consistency of the stool will be recorded at 6th week of intervention

SECONDARY OUTCOMES:
the number of stools delivered at 6th week of intervention | the number of the stools will be recorded at the 6th week of intervention
the number of incontinence episodes | the number of the incontinence episodes will be recorded at the 6th week of intervention
the number of painful defecation | the number of painful defecation will be recorded at the 6th week of intervention
the number of episodes of abdominal pain | the number of the episodes of abdominal pain will be recorded at the 6th week of intervention
the number of patients needed laxatives during treatment | the number patiens needed laxatives will be recorded for six weeks of intervention
side effects | the number and the character of the side effects will be recorded for six weeks of intervention
  the number and character of the sides effects will be recorded by the patient at the diary during the 6 weeks of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Horvath, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Dpt of Pediatrics The Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Dziechciarz P, Horvath A, Szajewska H. Polyethylene glycol 4000 for treatment of functional constipation in children. J Pediatr Gastroenterol Nutr. 2015 Jan;60(1):65-8. doi: 10.1097/MPG.0000000000000543. PMID 25162362